CLINICAL TRIAL: NCT06877728
Title: Comparative Effect of Neck Isometrics and Deep Cervical Flexion Exercises on Neck Pain, Functional Disability, Range of Motion and Muscle Weakness Among Breastfeeding Females
Brief Title: Comparative Effect of Neck Isometrics and Deep Cervical Flexion Exercises on Neck Pain Among Breastfeeding Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S23C14G92015
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain; Range of Motion; Muscle Weakness; Breastfeeding
Keywords: Neck pain; range of motion; Muscle weakness; Breastfeeding
MeSH Terms: conditions — Neck Pain; Muscle Weakness; Breast Feeding

STUDY DESIGN:
Intervention Model Description: participants received scar mobilization combined with kinesio tapping
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric exercises with conservative treatment (Active Comparator): Will receive Neck isometrics exercises with conservative treatment. Neck isometric exercises: 3 times weekly for 6 consecutive weeks (18 sessions) Duration: 10 to 15 repetitions with 3 sets, and 6 sec hold in flexion, extension and side flexion on both right and left.
  Interventions: Other: Neck isometric exercises: 3 times weekly for 6 consecutive weeks (18 sessions)
- Deep cervical flexion exercises with conservative treatment (Other): Will Deep cervical flexion exercises without conservative treatment. Deep cervical flexion exercises: 3 times weekly for 6 consecutive weeks (18 session) Duration: 10 to 15 repetitions with 3 sets, 30 sec rest given between each set. Exercise should target on deep cervical muscle rather than superficial muscle. Exercise should be conducted in supine position.
  Interventions: Other: Neck isometric exercises: 3 times weekly for 6 consecutive weeks (18 sessions)

INTERVENTIONS:
Other: Neck isometric exercises: 3 times weekly for 6 consecutive weeks (18 sessions) — Neck isometric exercises: 3 times weekly for 6 consecutive weeks (18 sessions) Duration: 10 to 15 repetitions with 3 sets, and 6 sec hold in flexion, extension and side flexion on both right and left.

SUMMARY:
Neck pain is a common complaint among breastfeeding females, potentially attributed to sustained postures and muscle imbalance. Breastfeeding females experiencing neck pain, aged between 18-40 years, will be recruited through local healthcare facilities and community outreach. The physical demands of breastfeeding, such as prolonged postures and repetitive movements, can contribute to the development of musculoskeletal issues in the cervical region.

Despite the prevalence of neck discomfort among breastfeeding females, there is a paucity of research exploring effective exercise interventions tailored to this specific population. Mothers' awareness of proper nursing positions during breastfeeding may have positive impact on the connection between mother and baby. Most typical positions for nursing a baby are cross cradle hold, cradle hold, side lying and football hold. Most common adapted breastfeeding position is cross cradle.

DETAILED DESCRIPTION:
A randomized control trial will be conducted to assess and compare the effectiveness of neck isometrics and deep cervical flexion exercises in alleviating neck pain, reducing disability, improving range of motion, and addressing muscle weakness in breastfeeding females. A sample size of 48 lactating women will be taken. Data will be collected from private clinical setups of Bahawalpur by using (NPRS) Numeric Pain Rating Scale Questionnaire, (NDI) Neck Disability Index, Range of motion will be assessed by inclinometer and Muscle strength will be assessed by MMT. A written consent form will be taken from participants meeting inclusion criteria and will be randomly allocated into two groups of equal members. Group A will be given Neck Isometric Exercises and Conservative treatment for 30 min (3-4days/week) of duration for total 6 weeks.

Group B will be given Deep Cervical Flexion Exercises with conservative treatment. The interventions will be provided for 30 minutes for 3-4 Day/week for 6 weeks. All participants in both groups will be evaluated before and after the treatment programs. Outcome measures will be calculated after 6 weeks of intervention. Data will be analyzed by using SPSS 21

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 25 to 40 years
* Mode of delivery (vaginal/c-section)
* Severe neck weakness (above grade III)
* Primigravida

Exclusion Criteria:

* Previous history of upper extremity musculoskeletal symptoms
* Radicular neck pain
* History of inflammatory disease (myelopathy)
* History of cervical fracture

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Breastfeeding females are included in the study.
Enrollment: 48 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
1. Numeric Pain Rating Scale (NPRS) | 8 Weeks
  A Numeric Pain Rating Scale (NPRS) is a commonly used self-report measure to assess pain intensity. It typically involves asking individuals to rate their pain on a numerical scale.
  Below is a suggested format for a Numeric Pain Rating Scale questionnaire along with instructions and scoring guidelines. Scoring: Ask participants to circle the number on the scale that corresponds to their current pain intensity. The score is a single numeric value ranging from 0 to 10, with 0 indicating no pain and 10 indicating the worst imaginable pain.
  The higher the score, the greater the perceived pain intensity. The NPRS is a widely used subjective pain measure that has good test-retest reliability (r=. 79-. 96)
NECK DISABILITY INDEX QUESTIONNARE | 8 Weeks
  The Neck Disability Index (NDI) is a widely used self-report questionnaire designed to assess disability related to neck pain. The questionnaire consists of 10 items that measure various aspects of daily activities affected by neck pain. Each item is scored on a 0 to 5 scale, and the total score is expressed as a percentage, with 0 indicating "no disability" and 5 indicating "complete disability. Format: 10 items evaluating concerns relating to neck pain.
  The participant selects the number that best describes their level of disability for each activity. The NDI has a fair to moderate test-retest reliability in patients with mechanical neck pain, intra class correlations can change between 0,50 and 0,98 (
INCLINOMETER NECK ROM: | 8 Weeks
  An inclinometer is a device used to measure the range of motion (ROM) of joints, including the neck, an inclinometer is often applied to measure flexion, extension, lateral flexion, and rotation of the cervical spine. The digital inclinometer demonstrated excellent reliability (ICC=0.75-0.86), except for the right lateral flexion (ICC=0.74) and left rotation (ICC=0.72)
MANUAL MUSCLE TESTING FOR MUSCLE WEAKNESS: | 8 Weeks
  Manual Muscle Testing (MMT) is a clinical and functional assessment technique used by healthcare professionals, such as physical therapists and physicians, to evaluate muscle strength and identify potential muscle weakness. It involves the application of resistance against a person's voluntary muscle contraction, and the resulting force is graded on a scale.
  5/5: Normal strength (complete range of motion against gravity with full resistance) 4/5: Good strength (complete range of motion against gravity with moderate resistance) 3/5: Fair strength (complete range of motion against gravity with no resistance) 2/5: Poor strength (partial range of motion against gravity) 1/5: Trace movement (a flicker or trace of movement, but no joint motion) 0/5: No movement (complete paralysis)(

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Taufiq, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No